CLINICAL TRIAL: NCT05817045
Title: A Randomized, Double-Blind, Sham Controlled, Stratified, Pivotal Efficacy and Safety Study of the EmitBio RD-X19 Treatment Device in Individuals 40 Years of Age and Older With Mild COVID-19 in the At-Home Setting
Brief Title: Evaluation of the RD-X19 Treatment Device in Individuals With Mild COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EmitBio Inc. (Industry)
Responsible Party: Sponsor
Organization: KNOWBio Inc. (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EB-P30-01
Record Dates: First submitted 2023-04-14; First posted 2023-04-18 (Actual); Results first posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Volunteers meeting all inclusion criteria and none of the exclusion criteria will be randomized to the RD-X19 treatment arm or the sham treatment arm within each cohort in a 1:1 ratio according to a fixed schedule via a permuted block design.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Active (Active Comparator): RD-X19 Active Device
  Investigational device that uses 32 J/cm2 of electromagnetic energy to target the oropharynx.
  Interventions: Device: RD-X19
- Sham (Sham Comparator): RD-X19 Sham Device
  Investigational device that uses safe electromagnetic energy to target the oropharynx but at energy levels with a lower inactivation potential against SARS-CoV2 in vitro.
  Interventions: Device: Sham

INTERVENTIONS:
Device: RD-X19 — Investigational device that uses safe electromagnetic energy to target the oropharynx.
  Arms: Active
Device: Sham — Investigational device that uses safe electromagnetic energy to target the oropharynx but at energy levels with a lower inactivation potential against SARS-CoV-2 in vitro.
  Arms: Sham

SUMMARY:
This is a randomized, double-blind, sham controlled, stratified, pivotal efficacy and safety study of the EmitBio RD-X19 treatment device in Individuals 40 Years of age and older with Mild COVID-19 in the at-home setting.

DETAILED DESCRIPTION:
This is a randomized, double-blind, sham controlled, stratified, pivotal efficacy and safety study of the EmitBio RD-X19 device in individuals age 40 and older with mild COVID-19 (as defined by NIH and FDA) in the at-home setting. Study subjects will self-administer treatment twice daily, 5 minutes per treatment for 7 consecutive days. Subjects will remain on study for a total of 14 study days (± 2 days) for treatment and follow-up. Neither study subject nor clinical trial personnel will be aware of the subject's treatment assignment. Clinical safety and efficacy outcomes will be assessed via self-assessed signs and symptoms (e-diary entries twice a day during the entire study period) with daily study staff checks, including home visits, and/or clinic visits for objective clinical assessments (vital signs, targeted physical exams, oropharyngeal exams) on study days 1, 5, 8 and 14.

The primary goal of the study is to evaluate the safety and efficacy of the RD-X19 treatment device to provide sufficient evidence to FDA to justify the authorization and/or approval of the device for treatment of subjects with mild COVID-19, age 40 and older in the home setting. Every attempt will be made to continue to follow safety in any study subject choosing to terminate the study early and all study subjects who progress to moderate or more severe forms of COVID-19 will be immediately referred for appropriate medical care. Medically necessary care of study participants will always take precedence over research.

ELIGIBILITY:
Inclusion Criteria:

1. Positive for SARS-CoV-2 as detected using an FDA authorized SARS-CoV-2 antigen test at the screening/baseline visit.
2. Negative for Influenza A and B antigen using an FDA-authorized rapid diagnostic test.
3. At least two moderate or greater COVID-19 signs and symptoms from the following list: cough, sore throat, nasal congestion, headache, chills and/or sweats, myalgia, fatigue, nausea (with or without vomiting) or one moderate or greater symptom and fever (temperature ≥ 100.5 degrees F).
4. Time from appearance of first COVID-19 sign or symptom to screening must be 72 hours or less.
5. Males or females, including pregnant and fecund females, 40 years of age and older on the date of enrollment.
6. BMI <40
7. Provides written informed consent prior to initiation of any study procedures.
8. Be able to understand and agrees to fully comply with defined and described study procedures and be available for all study visits for the entire study duration.
9. Agrees to collection of a nasopharyngeal swab for qPCR at baseline for the purposes of assessing viral burden as a potential covariate in data analyses and for genetic sequencing to characterize the predominant SARS-CoV-2 variants present in the study population.
10. Agrees to perform self-diagnostic home testing twice a day, separated by ≥ 6 hours for the entire length of the study.
11. Agrees to restrict medications used for symptomatic relief of signs and symptoms of COVID-19 during the study period, and, if used, to report ALL such medications (including home remedies) to the study staff.
12. Agrees to avoid the use of oral rinses and toothpastes containing alcohol-based compounds (e.g. Eucalyptol, Menthol, Thymol, Phenol) and/or Salicylates during the study period. Oral rinses, breath fresheners and toothpaste not containing these compounds are allowed.
13. Agrees to avoid nasal and sinus saline lavage during the study period.
14. No uncontrolled disease process (chronic or acute), other than COVID-19 signs and symptoms (See section 8.1.1 - General Screening)*.
15. No physical or mental conditions or attributes at the time of screening, which in the opinion of the PI, will prevent full adherence to, and completion of, the protocol.

Exclusion Criteria:

1. Positive for Influenza A and B antigen using an FDA-authorized rapid diagnostic test.
2. Individuals < age 40 on study day 1.
3. Individuals who are symptomatic for COVID-19 for more than 72 hours on study day 1.
4. COVID-19 signs associated with moderate or greater disease with evidence of lower respiratory involvement including shortness of breath (SOB) at rest or as determined by an exertional SOB protocol, SpO2 ≤94, respiratory rate ≥20 breaths per minute, heart rate ≥90 beats per minute, or abnormal pulmonary imaging.
5. Any medical disease or condition that, in the opinion of the site Principal Investigator (PI) or appropriate sub-investigator, precludes study participation.
6. History of use of a rescue inhaler for uncontrolled asthma within one month of study day 1.
7. History of recurrent alcohol intoxication or other recreational drug use (excluding medically prescribed cannabis) within one month of study day 1.
8. History of use, within one month of study day 1, of any FDA-authorized treatment for COVID-19. Use of non-approved putative therapies for COVID-19 (hyroxycholorquine, ivermectin, azithromycin) must be discontinued prior to enrollment in the study.
9. History of any systemic antiviral therapies within one month of study day 1.
10. History of oral or parenteral corticosteroid use within one month of study day 1. Active use of nasal or inhalable steroids is also exclusionary. Topical steroids are not exclusionary.
11. History of any chronic medical condition that has required adjustments to the type, dose or schedule of medical treatments within one month of study day 1.
12. Requirement to use narcotic medication for analgesia.
13. History of vasomotor rhinitis with or without post-nasal drip within one month of study day 1.
14. History of hypersensitivity or severe allergic reaction (e.g., anaphylaxis, generalized urticaria, angioedema, other significant reaction) to sun exposure.
15. Presence of any oral abnormality (e.g., including, but not limited to, ulcer, oral candidiasis, oral mucositis, symptomatic gingivitis, history of frequent recurrent aphthous ulcers, burning mouth syndrome, dry mouth syndrome, a disease that can result in xerostomia (e.g., Sjogren's syndrome), Temporomandibular Joint Syndrome, or other oral disorder that in the opinion of the investigator would interfere with device use and evaluation.
16. Any intra-oral metal body piercings that cannot be removed for the duration of the study. Metal orthodontia is permitted as braces will be covered by the device mouthpiece.
17. Any individual without teeth or with a dental malformation that precludes directed use of the device as intended.
18. Currently enrolled in or plans to participate in another clinical trial with a therapeutic investigational agent for any medical indication that will be received during the study period.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2023-04-21 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director EB-P30-01, Study Director — EmitBio
Locations (48):
- United States (48):
  - 322 - Desert Clinical Research/CCT Research, Mesa, Arizona
  - 347 - Velocity Clinical Research, Phoenix, Arizona
  - 312 - Smart Cures Clinical Research, Anaheim, California
  - 313 - Benchmark Southern California, Colton, California
  - 307 - Ark Clinical Research, Long Beach, California
  - 329 - Valley Clinical Trials, Northridge, California
  - 348 - San Francisco Research Institute, San Francisco, California
  - 328 - Mills Clinical Research, West Hollywood, California
  - 305 - Indago Research and Health Center, Hialeah, Florida
  - 321 - Helios Clinical Research - Kissimmee, Kissimmee, Florida
  - 310 - Accel Research Sites - St. Petersburg, Largo, Florida
  - 306 - Miami Clinical Research, Miami, Florida
  - 341 - Lifeline Primary Care / CCT Research, Lilburn, Georgia
  - 349 - Chicago Medical Research, Chicago, Illinois
  - 333 - Prime Global Research Inc., Chicago, Illinois
  - 331 - Chicago Clinical Research Institute, Chicago, Illinois
  - 345 - The Iowa Clinic/Avacare Legacy, West Des Moines, Iowa
  - 337 - Versailles Family Medicine/CCT Research, Versailles, Kentucky
  - 346 - Benchmark Research, Metairie, Louisiana
  - 323 - Annapolis Internal Medicine/CCT Research, Annapolis, Maryland
  - 324 - Advanced Primary and Geriatric Care / CCT Research, Rockville, Maryland
  - 327 - The Research Institute, Springfield, Massachusetts
  - 315 - Revival Research Institute - Dearborn, Dearborn, Michigan
  - 314 - Revival Research Institute - Sterling Heights, Sterling Heights, Michigan
  - 318 - Olive Branch Family Medical Center, Olive Branch, Mississippi
  - 335 - Clay Platte Family Medicine/CCT Research, Kansas City, Missouri
  - 336 - St. Louis Medical Professional/CCT Research, St Louis, Missouri
  - 344 - Skyline Medical Center/ CCT Research, Elkhorn, Nebraska
  - 326 - Healor Primary Care, Las Vegas, Nevada
  - 325 - Santa Rosa Medical Centers of Nevada / CCT Research, Las Vegas, Nevada
  - 302 - WellNow - East Amherst, East Amherst, New York
  - 316 - WellNow - Niskayuna, Niskayuna, New York
  - 332 - Prime Global Research Inc., The Bronx, New York
  - 338 - Carolina Internal Medicine Associates, Asheville, North Carolina
  - 320 - M3 Wake Research, Raleigh, North Carolina
  - 304 - WellNow - Cincinnati, Cincinnati, Ohio
  - 301 - WellNow - Columbus, Columbus, Ohio
  - 303 - WellNow - Huber Heights, Dayton, Ohio
  - 334 - Medical Care/CCT Research, Elizabethton, Tennessee
  - 308B - Kurr Research @ Complete Health Partners, Hendersonville, Tennessee
  - 308 - Kur Research @Complete Health Partners, Nashville, Tennessee
  - 330 - Clinical Trial Network, Houston, Texas
  - 319 - Helios Clinical Research - Keller, Keller, Texas
  - 309 - Tranquility Clinical Research, Webster, Texas
  - 340 - Premier Family Medical/CCT Research, American Fork, Utah
  - 343 - Cope Family Medicine/ CCT Research, Bountiful, Utah
  - 342 - Ogden Clinical, Grand View/CCT Research, Roy, Utah
  - 339 - Olympus Family Medicine/CCT, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active | Sham
Started | 162 | 168
Completed | 147 | 157
Not Completed | 15 | 11
Not completed — Protocol Violation | 0 | 3
Not completed — Withdrawal by Subject | 10 | 7
Not completed — Physician Decision | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Device Deficiency | 1 | 0
Not completed — System Error | 1 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): The Full Analysis Set (FAS) will consist of the set of randomized subjects, excluding: (i) subjects who were mis-randomized; and (ii) subject IDs corresponding to study participants that were re-randomized under a different subject ID.
Groups:
- Total: Total of all reporting groups
Arm/Group | Active | Sham | Total
Number analyzed (Participants) | 161 | 166 | 327
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.39 (8.793) | 55.56 (10.180) | 54.98 (9.526)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 105 | 204
  Male | 62 | 61 | 123
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 45 | 53 | 98
  Not Hispanic or Latino | 112 | 112 | 224
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 38 | 34 | 72
  White | 112 | 117 | 229
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 161 | 166 | 327
Body Mass Index (BMI) [Mean (Standard Deviation); unit: Kg/m^2] — Body Mass Index in Kg/m2
  Kg/m^2 | 28.9498 (5.01187) | 29.5443 (4.92951) | 29.2525 (4.97137)
Total Baseline Disease Severity Score [Mean (Standard Deviation); unit: units on a scale] — Each assessed COVID-19 symptom (cough, sore throat, nasal congestion, headache, chills and/or sweats, myalgia, fatigue, and nausea (with or without vomiting) will be rated on a 4-point scale from none (0) to severe (3). The baseline disease severity score is defined as the sum of the eight individual scores divided by eight. The total score ranges from 0-3 with higher numbers representing more severe symptoms.
  units on a scale | 1.4977 (0.46739) | 1.4571 (0.45741) | 1.4771 (0.46209)
COVID-19 vaccination status [Count of Participants; unit: Participants] — Prior COVID-19 vaccination (yes, no)
  Participants
    Yes | 122 | 118 | 240
    No | 38 | 45 | 83
    Missing | 1 | 3 | 4
Baseline Log10 nasopharyngeal viral load [Mean (Standard Deviation); unit: log 10 copies/mL] — Nasopharyngeal viral load numerical values (copies/mL) are recorded at baseline. For the viral load quantitation assay, the specified lower limit of quantification (LLOQ) and limit of detection (LOD) are both 5.0 x 102 copies/mL (which is 2.6990 on the Log10 scale) and the upper limit of quantification (ULOQ) is 5.0 x 108 copies/mL (which is 8.6990 on the Log10 scale).
  log 10 copies/mL | 6.2527 (1.44278) | 6.2655 (1.53496) | 6.2592 (1.48778)
SARS-CoV-2 antigen test type [Count of Participants; unit: Participants]
  Flowflex | 86 | 93 | 179
  BinaxNOW | 75 | 73 | 148
Randomization Stratum [Count of Participants; unit: Participants]
  Age 40-49, Disease Severity Score < 1.25 | 9 | 10 | 19
  Age 40-49, Disease Severity Score >= 1.25 | 44 | 45 | 89
  Age >= 50, Disease Severity Score < 1.25 | 35 | 35 | 70
  Age >= 50, Disease Severity Score >= 1.25 | 73 | 76 | 149
Hours at screening since onset of first COVID-19 sign or symptoms [Mean (Standard Deviation); unit: hours] | 43.9 (14.36) | 40.8 (15.09) | 42.3 (14.80)
Baseline Risk Factor Score [Count of Participants; unit: Participants] — Baseline Risk Factor Score (BRFS) is a numerical score that considers 12 individual risk factors for progression. Each individual risk factor contributes 0 to the BRFS if not present and contributes a value of either 1 or 2 (as specified in SAP) if the individual risk factor is present at baseline. The BRFS covariate will be capped at 6 in order to avoid the undue influence of a few subjects with a very high score provided that the proportion of subjects with BRFS >= 6 is no more than 0.10. Higher scores signify a greater number of risk factors are present.
  Participants
    0 | 100 | 109 | 209
    1 | 44 | 33 | 77
    2 | 14 | 19 | 33
    3 | 3 | 3 | 6
    4 | 0 | 2 | 2
    5 | 0 | 0 | 0
    6 | 0 | 0 | 0
    >6 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Sustained Resolution of COVID-19 Signs and Symptoms Without Subsequent Symptom Recurrence or Disease Progression (Until the End of the Study)
Description: Each of eight symptoms (cough, sore throat, nasal congestion, headache, chills and or sweats, myalgia, fatigue, and nausea (with or without vomiting)) will be rated on a 4-point scale from none (0) to severe (3). Time to sustained resolution of COVID-19 signs and symptoms as measured by the time (in hours) when all eight symptoms have been assessed by the subject as none (0) or mild (1) and all symptoms remain at or below 1 until study Day 14. Subjects that are hospitalized will be censored at 360 hours, which corresponds to the end of the time window for the day 14. A subject not satisfying case (i) or (ii), who takes nirmatrelvir/ritonavir or molnupiravir after initiating study treatment will be censored at the time that they first took this antiviral medication. Subjects not satisfying case (i), (ii), or (iii) will be censored at the last time that they have e-diary data recorded.
Time Frame: Baseline through Day 14
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 161 | 166
Participants | 107 | 120
Statistical Analysis 1: Comparison: Active vs Sham; NPANCOVA analysis for time to sustained resolution of COVID-19 signs and symptoms without subsequent recurrence or disease progression (until the end of the study) Full Analysis Set (FAS); Test type: Superiority — adjusted for the following prognostic baseline covariates: baseline log10 nasopharyngeal viral load, ethnicity, hours since symptom onset, and baseline risk factor score; p = 0.948, NPANCOVA; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.777 to 1.310] — For the HR calculation Sham was taken to be the reference group, meaning a HR > 1 is favorable for RD-X19
Statistical Analysis 2: Comparison: Active vs Sham; NPANCOVA analysis for time to sustained resolution of COVID-19 signs and symptoms without subsequent symptom recurrence or disease progression (until the end of the study) Per-Protocol Population; Test type: Superiority — Per-Protocol Population; p = 0.902, NPANCOVA — adjusted for the following prognostic baseline covariates: baseline log10 nasopharyngeal viral load, ethnicity, hours since symptom onset, and baseline risk factor score; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.774 to 1.337] — For the HR calculation Sham was taken to be the reference group, meaning a HR > 1 is favorable for RD-X19
Statistical Analysis 3: Comparison: Active vs Sham; NPANCOVA analysis for time to sustained resolution of COVID-19 signs and symptoms without subsequent symptom recurrence or disease progression (until the end of the study) - Secondary Analysis (FAS excluding subjects that were qPCR negative at baseline); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.859, NPANCOVA; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.782 to 1.342] — For the HR calculation Sham was taken to be the reference group, meaning a HR > 1 is favorable for RD-X19;

2. Primary Outcome: Kaplan-Meier Estimates for Time to Sustained Resolution of COVID-19 Signs and Symptoms Without Subsequent Symptom Recurrence or Disease Progression (Until the End of the Study) Full Analysis Set (FAS)
Description: Each of eight symptoms (cough, sore throat, nasal congestion, headache, chills and or sweats, myalgia, fatigue, and nausea (with or without vomiting)) will be rated on a 4-point scale from none (0) to severe (3). Time to sustained resolution of COVID-19 signs and symptoms as measured by the time (in hours) when all eight symptoms have been assessed by the subject as none (0) or mild (1) and all symptoms remain at or below 1 until study Day 14. Subjects that are hospitalized will be censored at 360 hours, which corresponds to the end of the time window for the day 14 visit. A subject not satisfying case (i) or (ii), who takes nirmatrelvir/ritonavir or molnupiravir after initiating study treatment will be censored at the time that they first took this antiviral medication. Subjects not satisfying case (i), (ii), or (iii) will be censored at the last time that they have e-diary data recorded.
Time Frame: Baseline through Day 14
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: hours
Arm/Group | Active | Sham
Number analyzed (Participants) | 161 | 166
hours
  25th percentile for time to sustained resolution: number analyzed (Participants) | 107 | 120
  25th percentile for time to sustained resolution | 44.22 [26.628 to 64.440] | 62.49 [41.338 to 70.551]
  Median time to sustained resolution: number analyzed (Participants) | 107 | 120
  Median time to sustained resolution | 100.36 [80.264 to 137.830] | 113.39 [89.617 to 140.690]
  75th percentile for time to sustained resolution: number analyzed (Participants) | 107 | 120
  75th percentile for time to sustained resolution | NA [209.970 to NA] — Subjects did not meet the 75th percentile | 261.35 [205.188 to NA] — Subjects did not meet the 75th percentile

3. Secondary Outcome: Number of Subjects With Two Negative SARS-CoV-2 Antigen Tests (With a Minimum Time Between Tests of Six Hours) Without Subsequent Virological Rebound During the Subject's Remaining Time on Study
Description: Number of subjects with two negative SARS-CoV-2 antigen tests (with a minimum time between tests of six hours) without subsequent virological rebound during the subject's remaining time on study. Subjects that are hospitalized will be censored at 360 hours, which corresponds to the end of the time window for the day 14 visit. A subject not satisfying case (i) or (ii), who takes nirmatrelvir/ritonavir or molnupiravir after initiating study treatment will be censored at the time that they first took this antiviral medication. Subjects not satisfying case (i), (ii), or (iii) will be censored at the last time that they have e-diary data recorded
Time Frame: Baseline through Day 14
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 161 | 166
Participants | 146 | 157
Statistical Analysis 1: Comparison: Active vs Sham; NPANCOVA analysis for time to first of two negative SARS-CoV-2 antigen tests (with a minimum time between tests of six hours) without subsequent virologic rebound (during the subject's remaining time on study) Full Analysis Set (FAS); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.017, NPANCOVA; Hazard Ratio (HR) = 1.29, 95% CI 2-sided [1.047 to 1.596] — For the HR calculation Sham was taken to be the reference group, meaning a HR > 1 is favorable for RD-X19
Statistical Analysis 2: Comparison: Active vs Sham; NPANCOVA analysis for time to first of two negative SARS-CoV-2 antigen tests (with a minimum time between tests of six hours) without subsequent virological rebound (during the subject's remaining time on study) (Per-Protocol population); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.014, NPANCOVA; Hazard Ratio (HR) = 1.33, 95% CI 2-sided [1.059 to 1.665] — For the HR calculation Sham was taken to be the reference group, meaning a HR > 1 is favorable for RD-X19;
Statistical Analysis 3: Comparison: Active vs Sham; NPANCOVA analysis for time to first of two negative SARS-CoV-2 antigen tests (with a minimum time between tests of six hours) without subsequent virological rebound (during the subject's remaining time on study) - Secondary analysis - (FAS excluding subjects that were qPCR negative at baseline); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.007, NPANCOVA; Hazard Ratio (HR) = 1.35, 95% CI 2-sided [1.086 to 1.690] — For the HR calculation Sham was taken to be the reference group, meaning a HR > 1 is favorable for RD-X19
Statistical Analysis 4: Comparison: Active vs Sham; Cox proportional hazards model for time to first of two negative SARS-CoV-2 antigen tests (with a minimum time between tests of six hours) without subsequent virological rebound (during the subject's remaining time on study) (FAS); Test type: Superiority — SARS-CoV-2 rapid antigen test type: Flowflex; Cox Proportional Hazard = 1.46, 95% CI 2-sided [1.064 to 1.997] — For the HR calculation Sham was taken to be the reference group, meaning a HR > 1 is favorable for RD-X19
Statistical Analysis 5: Comparison: Active vs Sham; Subgroup Analysis - Cox proportional hazards model for time to first of two negative SARS-CoV-2 antigen tests (with a minimum time between tests of six hours) without subsequent virological rebound (during the subject's remaining time on study) (FAS); Test type: Superiority — SARS-CoV-2 rapid antigen test type: BinaxNOW; Cox Proportional Hazard = 1.12, 95% CI 2-sided [0.801 to 1.561] — For the HR calculation Sham was taken to be the reference group, meaning a HR > 1 is favorable for RD-X19

4. Secondary Outcome: Kaplan-Meier Estimates Time to First of Two Negative SARS-CoV-2 Antigen Tests
Description: time to first of two negative SARS-CoV-2 antigen tests (with a minimum time between tests of six hours) without subsequent virologic rebound (during the subject's remaining time on study) Full Analysis Set (FAS)
Time Frame: Baseline through Day 14
Population: Full Analysis Set (FAS)
Measure: Number (95% Confidence Interval); unit: hours
Arm/Group | Active | Sham
Number analyzed (Participants) | 161 | 166
hours
  25th percentile for time to first of two negative SARS-CoV-2 tests: number analyzed (Participants) | 146 | 157
  25th percentile for time to first of two negative SARS-CoV-2 tests | 47.02 [41.241 to 60.457] | 52.89 [40.966 to 66.051]
  Median time to first of two negative SARS-CoV-2 tests: number analyzed (Participants) | 146 | 157
  Median time to first of two negative SARS-CoV-2 tests | 74.58 [70.741 to 87.604] | 87.97 [75.473 to 96.581]
  75th percentile for time to first of two negative SARS-CoV-2 tests: number analyzed (Participants) | 146 | 157
  75th percentile for time to first of two negative SARS-CoV-2 tests | 111.18 [100.228 to 121.916] | 133.42 [114.496 to 144.960]

5. Other Pre Specified Outcome: Secondary Qualitative Measures: COVID-19-related Assessment at Baseline, Day 5, 8 and 14/ET Visits (Full Analysis Set)
Description: The following are secondary qualitative measures (each taking the values yes, no) recorded at the post-baseline clinic visits for COVID-related assessment:
  In the past 24 hours, have you returned to your usual health (before your COVID-19 illness)? In the past 24 hours, have you returned to your usual activities (before your COVID-19 illness)?
Time Frame: Baseline, Day 5, Day 8, and Day 14 or Early Termination Visit
Population: Full Analysis Set (FAS)
Measure: Count of Participants; unit: Participants
Arm/Group | Active | Sham
Number analyzed (Participants) | 161 | 166
Participants
  Returned to usual health in past 24 hours (Day 5 visit): number analyzed (Participants) | 145 | 158
  Returned to usual health in past 24 hours (Day 5 visit): Yes | 48 | 48
  Returned to usual health in past 24 hours (Day 5 visit): No | 96 | 108
  Returned to usual health in past 24 hours (Day 5 visit): Missing | 1 | 2
  Returned to usual health in past 24 hours (Day 8 visit): number analyzed (Participants) | 147 | 158
  Returned to usual health in past 24 hours (Day 8 visit): Yes | 97 | 100
  Returned to usual health in past 24 hours (Day 8 visit): No | 46 | 54
  Returned to usual health in past 24 hours (Day 8 visit): Missing | 4 | 4
  Returned to usual health in past 24 hours (Day 14/ET visit): number analyzed (Participants) | 154 | 158
  Returned to usual health in past 24 hours (Day 14/ET visit): Yes | 129 | 132
  Returned to usual health in past 24 hours (Day 14/ET visit): No | 23 | 22
  Returned to usual health in past 24 hours (Day 14/ET visit): Missing | 2 | 4
  Returned to usual activities in past 24 hours (Day 5 visit): number analyzed (Participants) | 145 | 158
  Returned to usual activities in past 24 hours (Day 5 visit): Yes | 67 | 71
  Returned to usual activities in past 24 hours (Day 5 visit): No | 77 | 85
  Returned to usual activities in past 24 hours (Day 5 visit): Missing | 1 | 2
  Returned to usual activities in past 24 hours (Day 8 visit): number analyzed (Participants) | 147 | 158
  Returned to usual activities in past 24 hours (Day 8 visit): Yes | 115 | 115
  Returned to usual activities in past 24 hours (Day 8 visit): No | 28 | 38
  Returned to usual activities in past 24 hours (Day 8 visit): Missing | 4 | 5
  Returned to usual activities in past 24 hours (Day 14/ET visit): number analyzed (Participants) | 154 | 158
  Returned to usual activities in past 24 hours (Day 14/ET visit): Yes | 137 | 138
  Returned to usual activities in past 24 hours (Day 14/ET visit): No | 15 | 16
  Returned to usual activities in past 24 hours (Day 14/ET visit): Missing | 2 | 4

ADVERSE EVENTS:
Time Frame: 14 days
Description: Solicited and Unsolicited Treatment Emergent Adverse Events (TEAEs) will be recorded by clinical trial staff for the entire duration of the study, beginning after device administration and through day 14 or an early termination visit. No Adverse Events (AEs) that are not TEAEs are expected in this study since the time between enrollment and the first treatment is very brief. The safety population will consist of all randomized subjects who received any study treatment.
Arm/Group | Active | Sham
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/162
Serious Adverse Events (participants affected / at risk) | 0/158 | 0/162
Other Adverse Events (participants affected / at risk) | 18/158 | 12/162
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active (N=158) | Sham (N=162)
Headache (Nervous system disorders) | 4 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dry Mouth (Gastrointestinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Pharyngitis (Infections and infestations) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All study data and reports of study data are the property of the study sponsor. The sponsor may grant the PI the right to publish the results of this research in a scientific journal, conditional upon the review and concurrence of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/45/NCT05817045/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/45/NCT05817045/SAP_001.pdf